CLINICAL TRIAL: NCT01241136
Title: Open Wide Excision Versus Minimal Surgery for Pilonidal Disease: A Randomized Control Trial Evaluating for Early Recurrence and Patient Satisfaction
Brief Title: Open Wide Excision Versus Minimal Surgery for Pilonidal Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No recruitment occurred and the PI stopped the study.
Sponsor: United States Naval Medical Center, Portsmouth (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CIP# 10.0041
Record Dates: First submitted 2010-11-15; First posted 2010-11-16 (Estimated); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Pilonidal Disease
Keywords: pilonidal disease, cystectomy, recurrence
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Open traditional pilonidal cystectomy (Placebo Comparator): traditional complete wide-excision pilonidal cystectomy
  Interventions: Procedure: open wide-excision pilonidal cystectomy
- Minimal invasive pilonidal cystotomy (Experimental): Using only Keyes Trephines to unroof and curette the pilonidal cyst cavity
  Interventions: Procedure: minimal invasive pilonidal cystotomy

INTERVENTIONS:
Procedure: open wide-excision pilonidal cystectomy — traditional open wide-excisional pilonidal cystectomy
  Arms: Open traditional pilonidal cystectomy
Procedure: minimal invasive pilonidal cystotomy — unroofing the cyst cavity and curettage the cyst
  Arms: Minimal invasive pilonidal cystotomy

SUMMARY:
In order to compare the early recurrence rates of pilonidal disease and overall patient satisfaction between procedures involving minimal and wide open excisions, we propose to perform a prospective, randomized clinical trial comparing these two surgical procedures. Randomly assigned patients will undergo either 1) wide excisions of all pilonidal-diseased tissue (e.g. pits, cavity, sinus tracts), including a surrounding rim of normal tissue and left open to heal, or 2) minimal excisions of lined sinus tracts using varying sized trephines. Overall patient satisfaction will be evaluated by the amount of analgesic used for the procedure, the number of dressing changes, the length of convalescence, and overall patient tolerance of the procedures, both intra- and post-operatively. In addition, varying data points will be collected with the use of a quality of life survey and visual analog pain scale to analyze overall patient satisfaction. Patients will be followed for a period of two years following surgery to evaluate for early recurrence of their pilonidal disease.

DETAILED DESCRIPTION:
Pilonidal disease, a chronic infection involving the skin and subcutaneous tissues along the sacrococcygeal area (natal cleft) is a common disease affecting mostly young adult males who make up the majority of our military workforce. Surgical treatment options for pilonidal disease vary widely from the invasive (e.g. wide open excisions) to minimally invasive procedures (e.g. removal of lined sinus tracts using minimal excisions) as well as other popular treatments involving myocutaneous or skin flaps (Limberg flap and Z-plasty). All of these surgical procedures are associated with varying degrees of early and late recurrence rates; however, the current, more popular procedure for the treatment of pilonidal disease involves wide open excisions.

A recent advancement in the minimally invasive surgical technique for pilonidal disease involves the use of Keyes trephines (a 2-to-9 mm diameter biopsy instrument) to excise the individual pits and to drain the cyst cavities. Although this procedure has been proven to be effective against pilonidal disease with an overall low early recurrence rate, no clinical trial has been performed to rate this procedure of minimal excisions against the current, more common procedure of wide open excisions. A recent report has suggested that the recurrence rate of pilonidal disease for minimal excisions may be comparable to that of wide excisions. Furthermore, reports have also suggested that this minimally invasive procedure can be performed with minimal (and possibly local) anesthesia, less post-operative pain medication, and may involve a shorter convalescence time for patients.

In order to compare the early recurrence rates of pilonidal disease and overall patient satisfaction between procedures involving minimal and wide open excisions, we propose to perform a prospective, randomized clinical trial comparing these two surgical procedures. Randomly assigned patients will undergo either 1) wide excisions of all pilonidal-diseased tissue (e.g. pits, cavity, sinus tracts), including a surrounding rim of normal tissue and left open to heal, or 2) minimal excisions of lined sinus tracts using varying sized trephines. Overall patient satisfaction will be evaluated by the amount of analgesic used for the procedure, the number of dressing changes, the length of convalescence, and overall patient tolerance of the procedures, both intra- and post-operatively. In addition, varying data points will be collected with the use of a quality of life survey and visual analog pain scale to analyze overall patient satisfaction. Patients will be followed for a period of two years following surgery to evaluate for early recurrence of their pilonidal disease.

ELIGIBILITY:
Inclusion Criteria:

* All patients who are scheduled for elective surgical treatment for their pilonidal disease

Exclusion Criteria:

* 1. Any patient with active purulent infection (i.e. abscess). 2. Any patient who has had surgical intervention, excepting incisions and drainage for abscess for pilonidal disease.

Ages: 17 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-02-19 (Actual); Primary Completion 2014-11-25 (Actual); Study Completion 2025-07-16 (Actual)

PRIMARY OUTCOMES:
Rate of early recurrence | 2 years
  After surgical interventions, to see after 2 years the rate of recurrence of pilonidal disease

SECONDARY OUTCOMES:
Tolerance of the procedure | 30 days
  Determine wound healing times and amount of convalescence associated with each procedure
Patient satisfaction | 30 days
  Determine patient satisfaction factors using the quality of life survey and the post-operative visual analog pain scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Naval Medical Center Portsmouth, Portsmouth, Virginia, United States